CLINICAL TRIAL: NCT03687788
Title: The Effect of Laughter Therapy on Life Satisfaction and Loneliness in Older Adults Living in a Nursing Home: A Parallel Group Randomized Control Trial
Brief Title: The Effect of Laughter Therapy on Life Satisfaction and Loneliness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Pinar Zorba Bahceli, Asistant Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017/185
Record Dates: First submitted 2018-09-24; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Older Adults
Keywords: Laughter therapy; Loneliness; Life Satisfaction; Older adults; Nursing
MeSH Terms: conditions — Personal Satisfaction | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention group received laughter therapy twice a week for six weeks.
  Interventions: Behavioral: Laughter Therapy
- Control Group (No Intervention): The control group did not take part in the laughter therapy program. This group received the routine care given by the nurses in the center.

INTERVENTIONS:
Behavioral: Laughter Therapy — Laughter therapy program was composed of four steps. The first step, which took 10 minutes, had warm-up exercises including gentle stretching and hand clapping. The second step, which included deep breathing exercises and hand clapping, took 5 minutes. The third step involved children's games and laughter exercises. In this step, the most common laughter exercises were milkshake laughter, bugi bugi laughter techniques, lion laughter, cell phone, hot soup laughter, hug laughter, bird laughter, dialogue with nonsense, speech exercises, laugh at one's own aches and pains exercises, argument laughter, brushing teeth and mouthwash exercises. The sessions included a combination of different laughter exercises. This step took 15 minutes. The last step, which included wishes and resting by breathing, took 10 minutes.
  Arms: Intervention Group

SUMMARY:
Life satisfaction and loneliness are two important issues affecting the quality of life of the elderly. Older adults living in nursing homes experience the feeling of loneliness more and their life satisfaction decreases. For this reason, there is a need for an intervention that could increase the life satisfaction of the older adults and decrease their loneliness.

The aim of the research was to examine the effects of laughter therapy on life satisfaction and loneliness in older adults living in a nursing home.

DETAILED DESCRIPTION:
A single-blinded, parallel group randomized controlled trial was used to evaluate the impact of laughter therapy on life satisfaction and loneliness in older adults living in a nursing home.

The study was conducted in the only nursing home in Hatay province of Turkey.

The study participants were older adults living in a nursing home. A total of 62 older adults formed the experimental group (n = 31) and the control group (n = 31).

In order to ensure randomization and equal gender distribution, first, two groups (men and women) were formed. After the stratification process, five blocks consisting of six people and one group consisting of four people were formed using the permuted blocked randomization method. After the formation of the blocks, the elderly were randomly assigned to the experimental and the control group using a random number table. The experimental group received laughter therapy twice a week for 6 weeks and the usual care. The control group received only the usual care. To collect data, a personal information form, the De Jong Gierveld Loneliness Scale (DJGLS) and the Life Satisfaction Scale (LSS) were used.

ELIGIBILITY:
Inclusion Criteria:

* participants had to be 65 or older and be able to maintain independence in daily activities.

Exclusion Criteria:

* having severe hearing or perceptual deficits that impaired communication; having dementia, Alzheimer's disease, depression, uncontrolled diabetes, hypertensive disease and surgical operations with the risk of bleeding.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
De Jong Gierveld Loneliness Scale (DJGLS) scores | Change from Baseline De Jong Gierveld Loneliness Scale (DJGLS) scores at 6 weeks
  The De Jong Gierveld Loneliness Scale was originally developed by De Jong-Gierveld and Kamphuls (1985) and revised by De Jong Gierveld and Van Tilburg (1999). The 11-item DJGLS consists of two subscales: six negatively framed items measure emotional loneliness and five positively framed items measure social loneliness. The sum of these two subscales constitutes the general loneliness score. The scale is a Likert-type scale in which positive items are scored as 0 = yes, 1 = more or less, and 2 = no; and negative items are scored inversely as 2 = yes, 1 = more or less, and 0 = no. Total scores can range from 0 to 22, with a higher score denoting more severe loneliness. The DJGLS was tested for validity and reliability on Turkish population by Akgul and Yesilyaprak (2015), with Cronbach's alpha reliability coefficient of 0.85. In the present study, Cronbach's alpha was 0.87.

SECONDARY OUTCOMES:
Life Satisfaction Scale (LSS) scores | Change from Baseline Life Satisfaction Scale (LSS) scores at 6 weeks
  The Life Satisfaction Scale was developed by Diener et al. (1985). This five-point Likert scale, which has one factor structure, consists of 5 items and evaluates the life satisfaction of the individuals in general. The total score that could be obtained from the scale ranges from 5 to 25, and a higher scale score indicates a higher level of life satisfaction.
  The LSS was tested for validity and reliability within the Turkish population by Daglı and Baysal (2016), with Cronbach's alpha reliability coefficient of 0.88. In the present study, Cronbach's alpha was 0.89.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University Health Science Faculty, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuru Alici N, Zorba Bahceli P. Effects of Laughter Therapy on Life Satisfaction and Loneliness in Older Adults Living in Nursing Homes in Turkey: A Parallel Group Randomized Controlled Trial. Rehabil Nurs. 2021 Mar-Apr 01;46(2):104-112. doi: 10.1097/RNJ.0000000000000266. PMID 33646727